CLINICAL TRIAL: NCT01236625
Title: A Prospective Study on the Effect of Adhesiolysis During Elective Laparotomy or Laparoscopy on Per- and Postoperative Complication, Quality of Life and Socioeconomic Costs
Brief Title: The Effect of Adhesiolysis During Elective Abdominal Surgery on Per- and Postoperative Complication, Quality of Life and Socioeconomic Costs
Acronym: LAPAD
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RU-RTB-0003
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2010-09

CONDITIONS: Tissue Adhesions
Keywords: Tissue Adhesions; Adhesiolysis; Inadvertent enterotomy; Prospective cohort study; Quality of life
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No adhesiolysis: All patient undergoing elective laparotomy or laparoscopy with no need for adhesiolysis during the procedure.
- Adhesiolysis: All patient undergoing elective laparotomy or laparoscopy requiring adhesiolysis during the procedure.
  Interventions: Procedure: Adhesiolysis

INTERVENTIONS:
Procedure: Adhesiolysis — Blunt or sharp dissection of adhesive tissue.
  Groups: Adhesiolysis

SUMMARY:
Official title:

LAPAD - A prospective study on the effect of adhesiolysis during elective laparotomy or laparoscopy on per- and postoperative complication, quality of life and socioeconomic costs

Background:

With improved surgical technology and ageing of the population the number of reoperations in the abdomen dramatically increases. The risk for a repeat laparotomy or laparoscopy is a high as 30% in the first ten years after a laparotomy. In over 95% of reoperations adhesiolysis is required to gain access to the abdominal cavity and operation area. Adhesiolysis significantly increases the risk for inadvertent organ damage, such as enterotomies, leading to higher morbidity, mortality and socioeconomic costs.

Purpose:

To define the impact of adhesiolysis on per- and postoperative complications, quality of life and socioeconomic costs.

Design:

Prospective observational study.

Primary outcomes:

* adhesiolysis time
* inadvertent enterotomy
* seromuscular injury
* miscellaneous organ damage
* Serious adverse events of operation (anastomotic leakage, delayed diagnosed perforation, wound infection, abdominal infection, haemorrhage, pneumonia, urinary tract infection, abscess, fistula, sepsis, death)

Secondary outcomes:

* Hospital stay
* Intensive care admission
* Reinterventions
* In-hospital costs
* Parenteral feeding
* Short term readmissions (30 days)
* Quality of life (Gastro- intestinal tract complaints, Short Form- 36(SF-36), DASI (Duke Activity Score Index(DASI) )

Estimated enrollment: 800 start study: 1 june 2008 Inclusion completion date: 1 june 2010 Estimated study completion date: 1 february 2011

ELIGIBILITY:
Inclusion Criteria:

* Planned elective laparotomy or laparoscopy
* Mentally competent
* 18 years or older

Exclusion Criteria:

* Operation cancelled
* Bad quality of data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing elective laparotomy or laparoscopy in the department of surgery of the Radboud University Nijmegen Medical Centre (tertiary referral center).
Sampling Method: Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2008-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Inadvertent Enterotomy | Day of surgery (one day)
  Every unintended and iatrogenic full thickness defect of the bowel.
Seromuscular Injury | Day of surgery (one day)
  Every visible damage to the serosa, without leakage or exposure of the bowel lumen.
Miscellaneous Organ Damage | Day of surgery (one day)
  Unintended iatrogenic damage to intra- peritoneal organs and structures other than bowel. E.g. Spleen, liver, pancreas or ureter.
Serious Adverse Events | 30 days
  Complications marked as SAE: anastomotic leakage, delayed diagnosed perforation, wound infection, abdominal infection, haemorrhage, pneumonia, urinary tract infection, abscess, fistula, sepsis, death
Adhesiolysis Time | Day of surgery (one day)
  Time required to dissect adhesive tissue.

SECONDARY OUTCOMES:
Hospital stay | From surgery to discharge
  Number of days from surgery until discharge
Reinterventions | 30 days after discharge
  Emergency reoperation related to a complication of initial surgery within max. 30 days after discharge.
In- hospital Costs | From surgery to discharge
  Direct costs comprising costs from operation, stay on ward and Intesive Care Unit, medication use, diagnostics.
Parenteral Feeding | From surgery to discharge
  Number of days that patient required parenteral feeding.
Short term readmissions | 30 days after discharge
  Readmissions to the hospital related to complication of surgery.
Quality of life | 6 months post surgery
  Quality of life as measured with SF-36, Gastro- intestinal tract complaints and DASI index.

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, FRCS, Study Director — Radboud University Nijmegen Medical Center; Richard PG ten Broek, BsC, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] van Goor H. Consequences and complications of peritoneal adhesions. Colorectal Dis. 2007 Oct;9 Suppl 2:25-34. doi: 10.1111/j.1463-1318.2007.01358.x. PMID 17824967
- [Background] Van Der Krabben AA, Dijkstra FR, Nieuwenhuijzen M, Reijnen MM, Schaapveld M, Van Goor H. Morbidity and mortality of inadvertent enterotomy during adhesiotomy. Br J Surg. 2000 Apr;87(4):467-71. doi: 10.1046/j.1365-2168.2000.01394.x. PMID 10759744
- [Background] Parker MC, Ellis H, Moran BJ, Thompson JN, Wilson MS, Menzies D, McGuire A, Lower AM, Hawthorn RJ, O'Briena F, Buchan S, Crowe AM. Postoperative adhesions: ten-year follow-up of 12,584 patients undergoing lower abdominal surgery. Dis Colon Rectum. 2001 Jun;44(6):822-29; discussion 829-30. doi: 10.1007/BF02234701. PMID 11391142
- [Derived] Gawria L, Krielen P, Stommel MWJ, van Goor H, Ten Broek RPG. Reproducibility and predictive value of three grading systems for intraoperative adverse events in a cohort of abdominal surgery. Int J Surg. 2024 Jan 1;110(1):202-208. doi: 10.1097/JS9.0000000000000428. PMID 38000068
- [Derived] van den Beukel BAW, Toneman MK, van Veelen F, van Oud-Alblas MB, van Dongen K, Stommel MWJ, van Goor H, Ten Broek RPG. Elective adhesiolysis for chronic abdominal pain reduces long-term risk of adhesive small bowel obstruction. World J Emerg Surg. 2023 Jan 23;18(1):8. doi: 10.1186/s13017-023-00477-9. PMID 36691000
- [Derived] Strik C, Stommel MW, Schipper LJ, van Goor H, Ten Broek RP. Risk factors for future repeat abdominal surgery. Langenbecks Arch Surg. 2016 Sep;401(6):829-37. doi: 10.1007/s00423-016-1414-3. Epub 2016 Apr 13. PMID 27074725
- [Derived] Strik C, Stommel MW, Schipper LJ, van Goor H, Ten Broek RP. Long-term impact of adhesions on bowel obstruction. Surgery. 2016 May;159(5):1351-9. doi: 10.1016/j.surg.2015.11.016. Epub 2016 Jan 6. PMID 26767310
- [Derived] Strik C, ten Broek RP, van der Kolk M, van Goor H, Bonenkamp JJ. Health-related quality of life and hospital costs following esophageal resection: a prospective cohort study. World J Surg Oncol. 2015 Sep 4;13:266. doi: 10.1186/s12957-015-0678-3. PMID 26338109
- [Derived] Strik C, Stommel MW, Ten Broek RP, van Goor H. Adhesiolysis in Patients Undergoing a Repeat Median Laparotomy. Dis Colon Rectum. 2015 Aug;58(8):792-8. doi: 10.1097/DCR.0000000000000405. PMID 26163959
- [Derived] ten Broek RP, Strik C, van Goor H. Preoperative nomogram to predict risk of bowel injury during adhesiolysis. Br J Surg. 2014 May;101(6):720-7. doi: 10.1002/bjs.9479. PMID 24723023
- See also: main publication — http://www.ncbi.nlm.nih.gov/pubmed/23013804
- See also: publication as part of study — http://www.ncbi.nlm.nih.gov/pubmed/22791104